CLINICAL TRIAL: NCT05574127
Title: Brief Behavioral Activation for the Treatment of Depression in Older Adult Cancer Survivors
Brief Title: A Study of Brief Behavioral Activation for the Treatment of Depression in Older Adult Cancer Survivors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-248
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Survivorship
Keywords: Older Adult Cancer Survivors; history of cancer; 22-248; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Adult Cancer Survivors (OACS) - Behavioral Activation (BA) (Experimental): Older adult cancer survivors (OACS) will receive a Behavioral Activation intervention
  Interventions: Behavioral: Behavioral Activation
- Older Adult Cancer Survivors (OACS) - Supportive Psychotherapy (SP) (Experimental): Older adult cancer survivors (OACS) will receive a Supportive Psychotherapy intervention
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Behavioral Activation — Sessions for both arms (BP & SP) will be administered remotely via video-conference and/or telephone (per patient preference) at the following timeline:
  * Full participants (not training cases): Ten sessions (30-50 minutes each) will be delivered approximately weekly over a 10-week period (+10 weeks).
  * Training case participants: Ten sessions (30-50 minutes each) will be delivered over an approximately 5-week period (+10 weeks).
  Other Names: BA
  Arms: Older Adult Cancer Survivors (OACS) - Behavioral Activation (BA)
Behavioral: Supportive Psychotherapy — Sessions for both arms (BP & SP) will be administered remotely via video-conference and/or telephone (per patient preference) at the following timeline:
  * Full participants (not training cases): Ten sessions (30-50 minutes each) will be delivered approximately weekly over a 10-week period (+10 weeks).
  * Training case participants: Ten sessions (30-50 minutes each) will be delivered over an approximately 5-week period (+10 weeks).
  Other Names: SP
  Arms: Older Adult Cancer Survivors (OACS) - Supportive Psychotherapy (SP)

SUMMARY:
The purpose of this study is to find out if a psychotherapy method called behavioral activation (BA) can be successfully delivered by telephone or videoconference (remotely) and can effectively treat depression in Older Adult Cancer Survivors (OACS)

ELIGIBILITY:
Inclusion Criteria:

* As per self-report or medical record, ≥65 years old
* As per self-report or medical record, has a history of cancer
* As per medical record and/or clinician confirmation:

  * a patient in MSK Survivorship Clinics AND/OR
  * no evidence of disease (NED) AND/OR
  * 6 months or more post-treatment (patients on maintenance hormonal therapies are eligible)
* Fluent in English, as per self-reported fluency of "well" or "very well"*
* As per self-report, able to communicate over video-conference and/or phone for sessions
* Elevated score on the PHQ-9: ≥5 (N/A for Training Case participants)
* Received a Blessed Orientation-Memory-Concentration Scale (BOMC) score of ≤ 11 (N/A for Training Case participants)

Exclusion Criteria:

* As per PI determination, requires a higher level of care for current passive or active suicidal ideation than current protocol is able to provide. If a participant receives a score of > 0 on item 9 of the PHQ-9, they will be referred to study PI for further evaluation. They will be excluded from participation in this study if the PI determines they would be appropriate for a higher level of care than BA may be able to provide.
* As per self-report or as documented in the medical record, current untreated (e.g., no medication, no therapy) major psychotic disorder (schizotypal personality disorder, schizophreniform disorder, schizoaffective disorder). Patients diagnosed with a major psychiatric disorder will be reviewed by the study PI to determine eligibility prior to consent.
* As per self-report or medical record, currently taking antidepressant medication for < 3 month
* As per medical record, patient has impaired decision-making capacity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference of Patient Health Questionnaire 9 (PHQ-9) scores between study groups | 2 months post intervention
  Patient Health Questionnaire 9 (PHQ-9): The PHQ-9 consists of nine items, each of which corresponds to one of the nine symptoms required for a diagnosis of a major depressive disorder (MDD) as defined by the Diagnostic and Statistical Manual of Mental Disorders. Respondents are asked to rate how often they have been bothered by each of the nine symptoms over the preceding two weeks. Respondents rate each item on a four-point scale (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day). Its reliability and validity have been established in diverse general and medical populations. Total scores range from 0-27; In outpatient cancer settings, psychometric research suggests that a score of ≥8 indicates clinically significant depressive symptoms and should be used as a clinical cut-off .

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Saracino, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Saracino RM, Park EY, Demirjian C, Jutagir DR, McConnell KM, Schofield E, Raue PJ, Lejuez CW, Nelson CJ. Protocol for a randomized controlled trial of brief behavioral activation among older adult cancer survivors. J Geriatr Oncol. 2024 Jun;15(5):101719. doi: 10.1016/j.jgo.2024.101719. Epub 2024 Feb 10. PMID 38342735
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05574127/ICF_000.pdf